CLINICAL TRIAL: NCT05735821
Title: Comparison of Video and Breastfeeding Simulator Supported Training Activities for Mothers Who Couldn't Breastfeed Their Baby Staying in the Mother's Hotel
Brief Title: The Effectiveness of the Training Given to the Unable to Breastfeed Mothers Staying in the Mother's Hotel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HATİCE TETİK METİN (Other)
Collaborators: Atlas University (Other)
Responsible Party: Sponsor-Investigator, HATİCE TETİK METİN, Principal Investigator, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2022/043
Record Dates: First submitted 2022-12-28; First posted 2023-02-21 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Breast Feeding; Separation, Family
Keywords: Mother Hotel; Breastfeeding Education; Video and Breastfeeding Simulator; IMB Model; Maternal Attachment
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Trial model with randomized control, pretest-posttest control group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): The control group will be pre-tested with data collection tools and a post-test will be applied 1 month later. No intervention will be made.
- video group (Experimental): A pre-test will be applied to the video group. Afterwards, a video containing the breastfeeding education prepared by the researcher will be watched. A post-test will be administered after the training. After 1 month, contact will be made and the test will be done again.
  Interventions: Other: Giving breastfeeding training
- simulator group (Experimental): A pre-test will be applied to the simulator group. Afterwards, a training will be given by the researcher with a breastfeeding simulator. A final test will be given after the training. After 1 month, the contact will be made and the test will be done again.
  Interventions: Other: Giving breastfeeding training

INTERVENTIONS:
Other: Giving breastfeeding training — The control group will not be interfered with. Breastfeeding training will be given to the video and simulator group and the 3 groups will be compared.
  Arms: simulator group; video group

SUMMARY:
The study was planned as a randomized controlled study to evaluate the effectiveness of breastfeeding behavior development training using Video and Simulator, given to mothers whose babies are in the neonatal intensive care unit and who are staying in the mother's guesthouse.

As soon as the mothers who are separated from their babies and who have breastfeeding barriers come together with their babies and the breastfeeding barrier is lifted, to enable them to start breastfeeding effectively the effectiveness of the training, which will be given by applying 2 different methods based on the IMB (Knowledge, Motivation, Behavioral Skills) model will be evaluated.

The aim of the training is to develop breastfeeding behavior in mothers and to ensure a secure attachment between mother and baby.

(The research will be conducted in a randomized controlled trial model with a pretest-posttest control group.)

DETAILED DESCRIPTION:
The universe of the research; Bitlis State Hospital Newborn Unit will be formed by mothers whose babies are hospitalized and who stay at the mother's hotel.

Sample of the research:

G.Power 3.1.9.4 package program was used to calculate the sample size foreseen for the research. In the calculation made in this direction; sample size, 95% confidence interval, 0.6 effect value for 80% power was used, and it was seen that at least 90 individuals should be included in the study in total. Since the study will be conducted in 2 intervention and 1 control groups, it has been observed that there should be 30 people in each group.

Content of the Training Provided for Developing Breastfeeding Behavior Change; Training materials and training contents will be created by the researcher based on the IMB Model and the training will be planned. Trainings will be video supported and simulator supported. The video will be prepared by the researcher. The video will be prepared in accordance with the techniques of 'educational video development for e-Learning'. Breastfeeding Simulator will be tried to be obtained by applying to the Tübitak project. If Tübitak project support cannot be obtained, the Breastfeeding Simulator will be provided by the researcher.

Data collection stages: Participants who meet the sample selection criteria will be informed about the scope of the research and their verbal and written consent will be obtained.

Data Collection Tools

1. Socio-Demographic Data Questionnaire: The content will be created by the researcher by scanning the literature on the subject and in line with the suggestions of academicians specialized in Midwifery, Obstetrics and Gynecology Nursing.
2. Breastfeeding Self-Efficacy Scale
3. Maternal Attachment Scale
4. Knowledge levels and attitudes of mothers towards breastfeeding:The content will be created by the researcher by scanning the literature on the subject and in line with the suggestions of academicians specialized in Midwifery, Obstetrics and Gynecology Nursing.

The research will consist of 2 stages;

1. stage

The study will be started with the mothers in the control group. The mothers in the control group, who were selected in accordance with the sample selection criteria and agreed to be a participant, will be given data collection tools for the pre-test on the first day, and no intervention will be made other than the counseling given at the hospital. After 4 weeks from the pre-test, the mothers will be reached and the post-test will be applied.

Stage 2

The study will continue with the mothers in the Experimental group. Data collection tools will be applied to the mothers in the Experimental group, who were selected in accordance with the sample selection criteria and accepted to be a participant, for the pre-test on the first day to determine their levels. The training day will be planned for the mothers in the experimental group by determining the average length of stay of the babies. Training materials and training contents will be created by the researcher based on the IMB Model. The training period will be planned to last between 45 minutes and 1 hour. After the training, mothers will be given the opportunity to ask questions about the subjects they do not understand about the training given for 15 minutes and the training will be completed.

1. Experimental Group; The mothers in the 1st group will be pre-tested with data collection tools before the training, then video-assisted training will be given and the post-test will be applied after the training. After the mothers in this group are completed, the second group will be started.
2. Experimental Group; The mothers in the 2nd group will be pre-tested with the data collection tools before the training, then the Breastfeeding Simulator supported training will be given and the post-test will be applied after the training. Applications will be made to mothers participating in the training.

The retest of the two experimental groups will be applied 4 weeks after their training.

Statistical Analysis of Data

Analysis of the data will be done with SPSS 21.0 and will be studied at 95% confidence level. The kurtosis and skewness coefficients will be examined to determine the conformity of the variables to the normal distribution. It will be considered sufficient for the normal distribution that the kurtosis and skewness values obtained from the variables are between +3 and -3.

If normality is provided for the variables with skewness and kurtosis values between +3 and -3 obtained from the variables, parametric tests will be applied and non-parametric test techniques will be used for the variables outside this range. The independent groups t test for two groups, the examination of the variables providing normality in terms of variables with three or more groups, the ANOVA test, and the analysis of the variables that do not provide normality in terms of variables with three or more groups will be analyzed with the Kruskal test. In case of difference in ANOVA test, multiple comparisons will be analyzed with Tukey test and in Kruskal Wallis test with Mann Whitney test with bonferroni correction. Change will be analyzed by Iterative ANOVA test, in case of difference, multiple comparison dependent groups will be analyzed with t test. The relationship between categorical variables will be analyzed with the Chi-square test.

(NOTE: Consort Flow Chart will be followed)

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older,
* Mothers whose babies were admitted to the neonatal unit after delivery and stayed in the mother's guesthouse,
* Mothers of infants who did not breastfeed and bond within the first 30-60 minutes after birth and were immediately admitted to the newborn,
* Mothers who have not started breastfeeding their babies,
* Literate,
* Ability to understand and answer questions

Exclusion Criteria:

* Mothers whose babies were admitted to the neonatal unit after 24 hours
* Mothers who do not stay in the mother's guesthouse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
In education groups; Evaluation of personal data, obstetric data and newborn information with the Sociodemographic Data Questionnaire | at admission
  31 questions were created by the researcher by scanning the literature on the subject. The questions included women's socio-demographic characteristics, obstetric histories and newborn information.
In education groups; Measuring breastfeeding efficacy with the Breastfeeding Self-Efficacy Scale-Short Form | at admission
  The minimum score to be obtained from the breastfeeding self-efficacy scale is 14, and the maximum score is 70. A high score indicates high breastfeeding self-efficacy.
In education groups; Measuring the bond between mother and baby with the Maternal Attachment Scale | at admission
  The lowest score that can be obtained from the Maternal Attachment Scale is 26, and the highest score is 104. The Highest Score Indicates High Maternal Attachment.
In education groups; Determining the Percentage of the Number of Correct Answers to the Questions Regarding the Determination of Attitudes and Knowledge Levels towards Breastfeeding | at admission
  The questionnaire on Determining Attitudes and Knowledge Levels towards Breastfeeding consists of 14 questions.
In the control group; Evaluation of personal data, obstetric data and newborn information with the Sociodemographic Data Questionnaire | at admission
  31 questions were created by the researcher by scanning the literature on the subject. The questions included women's socio-demographic characteristics, obstetric histories and newborn information.
In the control group; Measuring breastfeeding efficacy with the Breastfeeding Self-Efficacy Scale-Short Form | at admission
  The minimum score to be obtained from the breastfeeding self-efficacy scale is 14, and the maximum score is 70. A high score indicates high breastfeeding self-efficacy.
In the control group; Measuring the bond between mother and baby with the Maternal Attachment Scale | at admission
  The lowest score that can be obtained from the Maternal Attachment Scale is 26, and the highest score is 104. The Highest Score Indicates High Maternal Attachment.
In the control group; Determining the Percentage of the Number of Correct Answers to the Questions Regarding the Determination of Attitudes and Knowledge Levels towards Breastfeeding | at admission,
  The questionnaire on Determining Attitudes and Knowledge Levels towards Breastfeeding consists of 14 questions.

SECONDARY OUTCOMES:
In education groups; Evaluation of Breastfeeding Efficiency with the Breastfeeding Self-Efficacy Scale-Short Form after the training given with the video and breastfeeding simulator | 1 week after training and 1 month after retraining
  The minimum score to be obtained from the breastfeeding self-efficacy scale is 14, and the maximum score is 70. A high score indicates high breastfeeding self-efficacy.
In education groups; Measuring the bond between mother and baby with the Mother Attachment Scale after the training given with the video and breastfeeding simulator | 1 week after training and 1 month after retraining
  The lowest score that can be obtained from the Maternal Attachment Scale is 26, and the highest score is 104. The Highest Score Indicates High Maternal Attachment.
In education groups; Determining the Rate of Correct Answers to the Questions Regarding the Determination of Attitudes and Knowledge Levels towards Breastfeeding after the training given with the video and breastfeeding simulator | 1 week after training and 1 month after retraining
  The questionnaire on Determining Attitudes and Knowledge Levels towards Breastfeeding consists of 14 questions.
In the control group; Measuring breastfeeding efficacy with the Breastfeeding Self-Efficacy Scale-Short Form | 1 month after entry
  The minimum score to be obtained from the breastfeeding self-efficacy scale is 14, and the maximum score is 70. A high score indicates high breastfeeding self-efficacy.
In the control group; Measuring the bond between mother and baby with the Maternal Attachment Scale | 1 month after entry
  The lowest score that can be obtained from the Maternal Attachment Scale is 26, and the highest score is 104. The Highest Score Indicates High Maternal Attachment.
In the control group; Determining the Percentage of the Number of Correct Answers to the Questions Regarding the Determination of Attitudes and Knowledge Levels towards Breastfeeding | 1 month after entry
  The questionnaire on Determining Attitudes and Knowledge Levels towards Breastfeeding consists of 14 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No